CLINICAL TRIAL: NCT01913873
Title: High-sensitivity Cardiac Troponin and CK-MB Concentrations in Patients Undergoing Cardiac Surgery
Brief Title: High-sensitivity Troponin in Cardiac Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Onze Lieve Vrouw Hospital (Other)
Collaborators: Roche Farma, S.A (Industry)
Responsible Party: Principal Investigator, Guy CAMMU, MD, PhD, Onze Lieve Vrouw Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: NATH201301
Record Dates: First submitted 2013-07-29; First posted 2013-08-01 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Heart; Dysfunction Postoperative, Cardiac Surgery; Myocardial Infarction; Myocardial Injury
Keywords: High-sensitivity Cardiac Troponin; Creatinin Kinase MB; Cardiac Surgery; Myocardial injury; Myocardial infarction; Concentration change
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cardiac biomarkers concentration changes (Experimental): In 2012 the Third Global MI Task Force has presented a third universal definition of MI implying that MI associated with CABG is arbitrarily defined by elevation of cardiac biomarkers values > 10x99th percentile URL in patients with normal baseline cTn values (≤ 99th percentile URL), in addition with either (i) new pathological Q waves or new LBBB (left bundle branch block), or (ii) angiographic documented new graft or new native coronary artery occlusion, or (iii) imaging evidence of new loss of viable myocardium or new regional wall motion abnormality.
  In this study we will measure the concentration changes over time of cardiac biomarkers (hs-cTN and CK-MB) and establish a threshold value for myocardial injury, diagnosed by ECG and approved -if necessary- by echocardiography.
  Interventions: Other: serum concentration changes cardiac biomarkers

INTERVENTIONS:
Other: serum concentration changes cardiac biomarkers — Serum concentration determination for cardiac biomarkers (CK-MB and Hs-cTn) preoperatively, at induction of anesthesia (after placement of the arterial line), upon arrival at the intensive care unit (ICU), as well as every 3 hours for 12 hours, then every 6 hours the following 12 hours and a last sample is taken 48 hours after surgery.

SUMMARY:
Among patients undergoing heart surgery, a measurable degree of heart muscle tissue injury is expected. The level of injury can be shown by measuring the blood levels of specific molecules called cardiac biomarkers. Those cardiac biomarkers are often used in the acute cardiac care to diagnose a myocardial infarction.

Postoperative heart infarction remains a frequent and important complication after heart surgery.Therefore it is important to recognize any cardiac event in patients who underwent heart surgery. Although different diagnostic tools can be used to recognize these events, few is known about the value of those cardiac biomarkers to diagnose a myocardial infarction after heart surgery.

In this study the investigators will describe the concentration changes of those cardiac biomarkers over time in patients undergoing heart surgery, and the investigators will try to establish a upper level value who could indicate heart infarction.

DETAILED DESCRIPTION:
This is a prospective interventional mono centre study. High-sensitivity troponin and CK-MB will be measured at different point of times in all adult patients undergoing cardiac surgery.

Experiments are conducted at the O.L.V. Hospital, Aalst, Belgium, in a fully equipped operating room and intensive care facility and in the presence of board-certified anesthesiologists for safety reasons. After approval by the institutional ethics committee and written informed consent, all adult patients scheduled for different types of cardiac surgery between June 2013 and June 2014 will be enrolled. Collected data include demographic information, presence of co-morbid conditions and basic preoperative laboratory testing (including Hs-cTn and CK-MB) (Table 1) as well as per- and postoperative factors (Table 2).

Four different surgeons will perform the surgeries. The revascularization strategy and work method are chosen according to each surgeon's preference and good clinical practice. Standard monitoring is used in all patients. Anaesthesia management is at the discretion of the attending anaesthesiologist and according to good clinical practice.

Serum levels of CK-MB and Hs-cTn will be measured at induction of anaesthesia (after placement of the arterial line), upon arrival at the intensive care unit (ICU), as well as every 3 hours for 12 hours, then every 6 hours the following 12 hours and a last sample is taken 48 hours after surgery. Samples are analysed at the department of Clinical Biochemistry of our institution with the Elecsys Troponin T hs immuno-assay. Lower limit of quantification being 0,14 Nano gram/L (company data).

Twelve-lead ECGs obtained routinely the day prior to surgery, immediately upon arrival at the ICU, and then 24 and 48 hours post-surgery will be retrospectively reviewed by a cardiologist blinded to all other data for evidence of new postoperative MI.

All cardiac events, as described by the Third Global MI Task Force definition of MI, will be noted. Additional ECG or transesophageal echocardiography will be done at the discretion of the attending ICU physician, according to ICU protocols and good clinical practice.

Approved automated record keeping system (MetaVision Suite, iMDSoft, the Netherlands) will be used in the ICU. The principal investigator and/or co-investigators will supervise data handling.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must be older than 18 years
* Undergoing cardiac surgery
* Each participant must have the mental capacity to decide whether he takes part in the trial or not.
* Each participant must voluntarily give his written informed consent.

Exclusion Criteria:

* Patients with severe or end-stage renal insufficiency.
* Insertion of assist devices.
* Surgery on urgent basis, that is, the same day after their coronary angiogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
high-sensitivity troponin T concentration changes over time in patients undergoing cardiac surgery | from 12 hours preoperatively to 48 hours postoperatively
  Serum levels of Hs-cTn (high-sensitivity cardiac troponin assays) will be measured from 12 hours preoperatively, at induction of anesthesia (after placement of the arterial line), upon arrival at the intensive care unit (ICU), as well as every 3 hours for 12 hours, then every 6 hours the following 12 hours and a last sample is taken 48 hours after surgery.
CK-MB concentration changes over time in patients undergoing cardiac surgery | From 12 hours preoperatively to 48 hours postoperatively
  Serum levels of CK-MB will be measured 12 hours preoperatively, at induction of anesthesia (after placement of the arterial line), upon arrival at the intensive care unit (ICU), as well as every 3 hours for 12 hours, then every 6 hours the following 12 hours and a last sample is taken 48 hours after surgery.

SECONDARY OUTCOMES:
Determination of threshold values for high-sensitivity troponin T and CK-MB cardiac biomarkers that strongly suggest substantial myocardial damage and necrosis. | every 3 postoperative hours for the first 12 hours, then every 6 hours the following 12 hours and a last sample is taken 48 hours after surgery
  Postoperative myocardial infarction remains a frequent and important complication after cardiac surgery. In 2012 the Third Global MI Task Force has presented a third universal definition of myocardial infarction (MI) implying that MI associated with coronary artery bypass grafting (CABG) is arbitrarily defined by elevation of cardiac biomarkers values > 10x99th percentile URL in patients with normal baseline cTn values (≤ 99th percentile URL), in addition with either (i) new pathological Q waves or new LBBB (left bundle branch block), or (ii) angiographic documented new graft or new native coronary artery occlusion, or (iii) imaging evidence of new loss of viable myocardium or new regional wall motion abnormality. Although some suggest that ECG, myocardial scan, and CK-MB criteria underestimate the prevalence of MI after CABG, few is known about the established threshold values for hs-cTn after valve surgery or combined surgery.

OTHER OUTCOMES:
Twelve-lead Electrocardiographs (ECGs) | the day prior to surgery, immediately upon arrival at the ICU, and then 24 and 48 hours post-surgery
  Twelve-lead ECGs obtained routinely will be retrospectively reviewed by a cardiologist blinded to all other data for evidence of new postoperative MI.

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie De Mey, MD, Principal Investigator — OLV Hospital Aalst, Belgium; Koen De Decker, MD, Principal Investigator — OLV Hospital Aalst, Belgium; Guy Cammu, MD,PhD, Principal Investigator — OLV Hospital Aalst, Belgium; Inger Brandt, MD, Study Chair — OLV Hospital Aalst, Belgium; Pierre Couture, MD, Study Chair — Montreal Heart Institute, Quebec, Canada; William Wijns, MD, Study Chair — OLV Hospital Aalst, Belgium; Jan Verbeke, MD, Study Chair — OLV Hospital Aalst, Belgium; Ivan Degrieck, MD, Study Chair — OLV Hospital Aalst, Belgium
Locations (1):
- Intensive Care Unit, OLV Hospital Aalst, Belgium, Aalst, East-Flanders, Belgium

REFERENCES:
- [Background] Thygesen K, Mair J, Katus H, Plebani M, Venge P, Collinson P, Lindahl B, Giannitsis E, Hasin Y, Galvani M, Tubaro M, Alpert JS, Biasucci LM, Koenig W, Mueller C, Huber K, Hamm C, Jaffe AS; Study Group on Biomarkers in Cardiology of the ESC Working Group on Acute Cardiac Care. Recommendations for the use of cardiac troponin measurement in acute cardiac care. Eur Heart J. 2010 Sep;31(18):2197-204. doi: 10.1093/eurheartj/ehq251. Epub 2010 Aug 3. PMID 20685679
- [Background] Morrow DA, Cannon CP, Jesse RL, Newby LK, Ravkilde J, Storrow AB, Wu AH, Christenson RH; National Academy of Clinical Biochemistry. National Academy of Clinical Biochemistry Laboratory Medicine Practice Guidelines: Clinical characteristics and utilization of biochemical markers in acute coronary syndromes. Circulation. 2007 Apr 3;115(13):e356-75. doi: 10.1161/CIRCULATIONAHA.107.182882. Epub 2007 Mar 23. No abstract available. PMID 17384331
- [Background] Apple FS, Jesse RL, Newby LK, Wu AH, Christenson RH; National Academy of Clinical Biochemistry; IFCC Committee for Standardization of Markers of Cardiac Damage. National Academy of Clinical Biochemistry and IFCC Committee for Standardization of Markers of Cardiac Damage Laboratory Medicine Practice Guidelines: Analytical issues for biochemical markers of acute coronary syndromes. Circulation. 2007 Apr 3;115(13):e352-5. doi: 10.1161/CIRCULATIONAHA.107.182881. Epub 2007 Mar 23. No abstract available. PMID 17384332
- [Background] Carrier M, Pellerin M, Perrault LP, Solymoss BC, Pelletier LC. Troponin levels in patients with myocardial infarction after coronary artery bypass grafting. Ann Thorac Surg. 2000 Feb;69(2):435-40. doi: 10.1016/s0003-4975(99)01294-1. PMID 10735677
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Writing Group on the Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Thygesen K, Alpert JS, White HD, Jaffe AS, Katus HA, Apple FS, Lindahl B, Morrow DA, Chaitman BA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S; ESC Committee for Practice Guidelines (CPG). Third universal definition of myocardial infarction. Eur Heart J. 2012 Oct;33(20):2551-67. doi: 10.1093/eurheartj/ehs184. Epub 2012 Aug 24. No abstract available. PMID 22922414
- [Background] Selvanayagam JB, Petersen SE, Francis JM, Robson MD, Kardos A, Neubauer S, Taggart DP. Effects of off-pump versus on-pump coronary surgery on reversible and irreversible myocardial injury: a randomized trial using cardiovascular magnetic resonance imaging and biochemical markers. Circulation. 2004 Jan 27;109(3):345-50. doi: 10.1161/01.CIR.0000109489.71945.BD. Epub 2004 Jan 19. PMID 14732755